CLINICAL TRIAL: NCT05393414
Title: Efficacy of NSAID and Acetaminophen in the Control of Post-Operative Pain in Patients Undergoing Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B0110219
Record Dates: First submitted 2022-05-13; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Pain; Hispanics; Opioid Use; Multimodal Analgesia; Total Knee Arthroplasty
Keywords: Total Knee Arthroplasty; Postoperative Pain; Opioid Use; Hispanics; Clinical Outcomes; Multimodal Analgesia
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Morphine; oxycodone-acetaminophen; Ketorolac; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid Sparing Multimodal Regimen (Experimental): After surgery, the experimental group will receive a combination of ketorolac 30 mg intravenous (IV) every six hours for patients younger than 65 years old or ketorolac 15mg IV every six hours for those older than 65 years old; and acetaminophen 1 gram by mouth (PO) every six hours up to 72 hours
  Interventions: Drug: Opioid sparing protocol
- Opioid Based Multimodal Regimen (Experimental): After surgery, the control group will receive a combination of morphine 0.1 mg/kg IV every six hours and oxycodone combined with acetaminophen (2.5 mg / 325 mg) two tabs PO every six hours up to 72 hours
  Interventions: Drug: Opioid based protocol

INTERVENTIONS:
Drug: Opioid based protocol — Use of combination of drug dosage frequency and duration of morphine injection with percocet oral as standard postoperative pain control for up to 72 hours as requested by each patient
  Other Names: morphine injection; percocet oral
  Arms: Opioid Based Multimodal Regimen
Drug: Opioid sparing protocol — Use of combination of drug dosage frequency and duration of ketorolac injection with acetaminophen oral as standard postoperative pain control for up to 72 hours as requested by each patient
  Other Names: ketorolac injection; acetaminophen oral
  Arms: Opioid Sparing Multimodal Regimen

SUMMARY:
An alternate perioperative pain control protocol composed of intravenous ketorolac and oral acetaminophen for patients who underwent total knee replacement was designed with the aim to determine its efficacy when compared to pain control with intravenous morphine and oral oxycodone combined with acetaminophen. In addition, the study will evaluate the differences and similarities in the Hispanic population that could predict protocol efficacy.

DETAILED DESCRIPTION:
Acute pain after a surgical procedure may occur secondary to trauma from the procedure itself or from procedure-related complications. Appropriate peri-operative acute pain management is an important phase of patient's recovery since it's under-treatment can lead to adverse outcomes such as: thromboembolic and pulmonary complications, additional time spent in an intensive care unit or hospital, hospital readmission for further pain management, needless suffering, impairment of health-related quality of life, and development of chronic pain. Furthermore, it's over-treatment with opioid medications is associated with an increased risk of thromboembolic, infectious and gastrointestinal complications as well as increased length of hospital stay, cost of care and risk of opioid addiction.

Perioperative administration of intravenous (IV) non steroidal anti-inflammatory drugs (NSAID), such as ketorolac, has been shown to effectively decrease opioid requirements and pain levels while demonstrating tolerable side effects. Its use after total knee replacement has been associated with a 27% decrease in the use of morphine. When NSAID is combined with acetaminophen 1000mg every six hours, an additional benefit in terms of improved pain scores on post-operative day three was shown in patients who underwent total hip or knee arthroplasty. Therefore, the purpose of this study is to provide an effective alternative for pain management in Hispanic patients who underwent total knee replacement and evaluate the role of ketorolac and acetaminophen.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic American patients undergoing primary total knee arthroplasty
* Older than 21 years of age
* Classified with an American Society of Anesthesiologist Classification (ASA) of I or II.

Exclusion Criteria:

* Hypersensitivity to any components of analgesic drugs
* Impaired renal, cardiac, or hepatic function
* Baseline serum creatinine level higher than 1.2mg/dL
* History of gastrointestinal bleeding
* Neuromuscular deformities
* Inability to consent

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Pain scores using numerical rating scale (NRS, 0 to 10) | Post-operative 12 hours after surgery
  The amount of pain intensity reported will be measure throughout the numerical rating scale. Each patient will rate their pain intensity on a scale from 0 to 10, where zero represents "no pain," whereas 10 represents the "most intense pain" (e.g., "the most intense pain imaginable," "the maximum pain intensity as it could be"); during the 12 hours postoperative period
Pain scores using numerical rating scale (NRS, 0 to 10) | Post-operative 24 hours after surgery
  The amount of pain intensity reported will be measure throughout the numerical rating scale. Each patient will rate their pain intensity on a scale from 0 to 10, where zero represents "no pain," whereas 10 represents the "most intense pain" (e.g., "the most intense pain imaginable," "the maximum pain intensity as it could be"); during the 24 hours postoperative period
Pain scores using numerical rating scale (NRS, 0 to 10) | Post-operative 48 hours after surgery
  The amount of pain intensity reported will be measure throughout the numerical rating scale. Each patient will rate their pain intensity on a scale from 0 to 10, where zero represents "no pain," whereas 10 represents the "most intense pain" (e.g., "the most intense pain imaginable," "the maximum pain intensity as it could be"); during the 48 hours postoperative period

SECONDARY OUTCOMES:
Hospital Length of Stay | up to 30 days
  The number of days per patient from the time of admission to discharge up to 30 days
Drug-related adverse events | From the time of surgery after being discharge (0 to 72 hours after surgery)
  nausea, dizziness, vomit, tachycardia, pruritus and headache

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Otero-Lopez, MD, Principal Investigator — Orthopaedic Surgery Section, University of Puerto Rico Medical Sciences Campus San Juan, Puerto Rico
Locations (1):
- University of Puerto Rico Medical Sciences Campus, Ortopaedic Surgery Department, San Juan, Puerto Rico